CLINICAL TRIAL: NCT01153334
Title: Efficacy of Early Intensive ROsuvastatin Therapy in Patients With ST-segment Elevation Myocardial Infarction Undergoing PrimARY Percutaneous Coronary Intervention (the ROSEMARY Trial)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2009-0277
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: ST-segment Elevation AMI

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early intensive rosuvastatin therapy (Experimental)
  Interventions: Drug: Early intensive rosuvastatin therapy (40 mg for 7days, starting in ER prior to primary PCI)
- Conventional statin therapy (Placebo Comparator)
  Interventions: Drug: Early intensive rosuvastatin therapy (40 mg for 7days, starting in ER prior to primary PCI)

INTERVENTIONS:
Drug: Early intensive rosuvastatin therapy (40 mg for 7days, starting in ER prior to primary PCI) — 1. Test group: Early intensive rosuvastatin therapy - rosuvastatin 40 mg for pre-PCI loading and 7 days post PCI and 10 mg daily thereafter 2. Control group: Conventional statin therapy - Placebo for pre-PCI loading in ER and rosuvastatin 10 mg daily after primary PCI

SUMMARY:
Objectives: An investigator-initiated, double-blind, randomized, placebo-controlled, multi-center study to evaluate the efficacy of early intensive rosuvastatin therapy (rosuvastatin 40 mg for pre-PCI loading and 7 days post PCI and 10 mg daily thereafter) versus low dose conventional statin therapy (placebo for pre-PCI loading and rosuvastatin 10 mg daily after primary PCI) on infarct size measured by cardiac MRI and clinical outcomes in STEMI patients undergoing primary percutaneous coronary intervention (PCI). Hypothesis: The infarct size in the early high dose rosuvastatin group is smaller than that of the control patients treated with low does conventional statin therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient had the symptoms of acute myocardial infarction within 12 hours with ST-segment elevation of more than 1 mm in at least two contiguous leads of EKG or new onset LBBB.
2. Male or female over 20 years of age
3. Signed written informed consent to participate in the study

Exclusion Criteria:

1. Congestive heart failure (NYHA Class III or IV) or LVEF <35%.
2. Clinically significant heart disease requiring CABG, cardiac transplantation, surgical repair and/or replacement during the course of the study.
3. Previous MI or CABG
4. Known serious or hypersensitivity reactions to statin, antiplatelet agents (aspirin or clopidogrel), or heparin.
5. Known familial hypercholesterolemia
6. Known skeletal muscle disease
7. Known active liver disease such as hepatitis or liver cirrhosis (except for fatty liver)
8. Renal failure (Cr >2.0 mg/dL)
9. Secondary causes of hyperlipoproteinemia: uncontrolled primary hypothyroidism, and/or nephrotic syndrome
10. Non-cardiac comorbidity with a life expectation < 1 year
11. Contraindications to CMRI (eg, implanted pacemaker or cardiac defibrillator, claustrophobia, etc.)
12. Pregnant or lactating women or women of childbearing potential
13. Participation in any investigational drug or device study within 30 days prior to study entry

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2010-08-02 (Actual); Primary Completion 2013-06-27 (Actual); Study Completion 2013-06-27 (Actual)

PRIMARY OUTCOMES:
Infarct size measured by cardiac MRI | day 3-7

CONTACTS AND LOCATIONS:
Overall Officials: Yangsoo Jang, M.D, Ph.D, Principal Investigator — Division of Cardiology, Severance Cardiovascular Hospital, Yonsei University Health System
Locations (1):
- Severance Hospital, Seoul, South Korea